CLINICAL TRIAL: NCT03490526
Title: Comparison Between Two Different Techniques of Root Canal Disinfection (XP-endo Finisher Versus Passive Ultrasonic Irrigation): Randomized Clinical Trial
Brief Title: Root Canal Disinfection: a Comparison Between Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO0024
Record Dates: First submitted 2018-03-15; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal disinfection with XP-endo Finisher (Experimental)
  Interventions: Device: Root canal disinfection with XP-endo Finisher
- Root canal disinfection with passive ultrasonic irrigation (Active Comparator)
  Interventions: Device: Root canal disinfection with passive ultrasonic irrigation

INTERVENTIONS:
Device: Root canal disinfection with XP-endo Finisher — The XP-Endo® finisher will be used next to the X-Smart Plus endodontic motor, with speed settings at 800rpm and torque at 1 N.cm. Irrigation with 17% EDTA and 2.5% NaOCl will be performed in three cycles of one minute each. In each cycle the XP-Endo will be used in the working length in continuous and slow movements of entrance and exit, with amplitude of 5mm, for a period of 1 minute, followed by new irrigation with 2.5ml of EDTA solution or hypochlorite of sodium 2,5%. Finally, the channel will be completely dry with absorbent paper tips
  Arms: Root canal disinfection with XP-endo Finisher
Device: Root canal disinfection with passive ultrasonic irrigation — For cleaning using passive ultrasonic irrigation, the E1 Irrisonic tip (Helse Ultrasonic, Ribeirão Preto, SP), will be used with Jetlaxis Sonic BP LED (Schuster, Santa Maria, RS). The insert has a diameter equivalent to a manual file 20, with reduced taper (0.01). The power used will be 10%. With root canals flooded with 17% EDTA, the irrigation tips will be coupled to the ultrasound and 1mm shorter than the working length. These tips will be kept in the center of the canal avoiding contact with the dentin walls. The irrigation will be performed in three cycles, and in each cycle the irrigation tips will be activated for 1 minute followed by new irrigation with 2.5ml EDTA. The same procedure will be repeated with 2.5% NaoCl. Finally, the channel will be completely dry with absorbent paper tips.
  Arms: Root canal disinfection with passive ultrasonic irrigation

SUMMARY:
Caries disease is still the leading cause of severe tooth decay. Since this can lead to tooth loss, it is important that appropriate treatment is advised to help prevent damage and maintain tooth health. Faced with major coronary destruction, several times it becomes necessary to perform the endodontic treatment, aiming to maintain the element in the buccal cavity for longer. It is known that an excellent restorative treatment with poor endodontic treatment and vice versa has a direct impact on the (in) success of the treatment. In this context, the proper cleaning of the root canals is highlighted, aiming the removal of bacteria and toxins. There are several cleaning methods described in the literature, but it is not yet known which would be the most effective in the removal of these contaminants. In this double-blind randomized clinical trial, patients who need and meet the inclusion criteria will undergo endodontic treatment in two different root canal cleansing techniques (passive ultrasonic cleaning and cleaning with the XP Endo device). Patients will be monitored annually after finish your endodontic treatment to evaluate the periradicular repair and the quality of endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more;
* good general healthy;
* molars or premolar requiring endodontic treatment;
* at least 20 teeth;

Exclusion Criteria:

* root fracture;
* injury involving the furcation region
* need to behave as a prosthetic abutment;
* mobility greater than degree I;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-02 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Periradicular repair | 2 years
  This outcome will be evaluated radiographically by one calibrated examiner.

SECONDARY OUTCOMES:
Quality of endodontic treatment | 2 years
  This outcome will be evaluated through a radiograph by one calibrated examiner.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No